CLINICAL TRIAL: NCT05186415
Title: Contrast Enhanced Three Dimensional Echocardiographic Quantification of Right Ventricular Volumes in Repaired Congenital Heart Disease
Brief Title: Contrast Enhanced 3D Echocardiographic Quantification of Right Ventricular Volumes in Repaired CHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Shannon N. Nees, MD, Pediatric Cardiologist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1764041-1
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Tetralogy of Fallot; Pulmonary Insufficiency
Keywords: ultrasound enhancing agent; echocardiography; lumason
MeSH Terms: conditions — Tetralogy of Fallot; Respiratory Insufficiency | interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- diagnostic arm (Experimental): Contrast enhanced 3D echo (Lumason)
  Interventions: Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Injection Powder for Suspension [LUMASON]

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Injection Powder for Suspension [LUMASON] — The patient will receive the weight-based dose of Lumason of 0.03 mL/kg per injection, not to exceed 2.4 mL per injection per the FDA and manufacturer recommendations.

SUMMARY:
We propose the novel integration of two echocardiographic technologies - three-dimensional echocardiography using semi-automated right ventricular analysis coupled with the administration of ultrasound enhancing agents - to improve the inter-rater reliability and accuracy of various measures of right ventricular size and function, compared with cardiac MRI.

DETAILED DESCRIPTION:
Patients with repaired congenital heart disease with residual pulmonary insufficiency represent a challenging group of patients with congenital heart disease as they develop progressive right ventricular dilation and failure, increasing the risk for sudden cardiac death and often necessitating pulmonary valve replacement. These patients require close follow-up with serial cardiac imaging; however, the complex three-dimensional structure of these dilated right ventricles renders them difficult to adequately image with traditional two-dimensional echocardiography. Due to these difficulties, cardiac MRI is the current gold standard for assessing right ventricular size and function in these patients. However, cardiac MRI is costly and less accessible for patients than echocardiography. Although initial studies comparing 3D echocardiography with MRI showed that 3D echocardiography underestimates right ventricular size, recent advances in three-dimensional imaging technologies which utilize automated ultrasound "speckle-tracking" and artificial intelligence technology are lessening this inherent bias. Furthermore, the use of commercially-available ultrasound enhancing agents made of lipid microspheres has improved left ventricular endocardial border detection, inter-rater reliability and correlation of 3D echocardiography obtained estimates of left ventricular size and function compared with Cardiac Magnetic Resonance (CMR). However, their use has yet to be applied to the three-dimensional echocardiographic assessment of the right ventricle in congenital heart disease despite their ability to improve right ventricular endocardial border detection with three-dimensional echocardiography in adults. The investigators propose the novel integration of two echocardiographic technologies - three-dimensional echocardiography using semi-automated right ventricular analysis coupled with the administration of ultrasound enhancing agents - to change the paradigm of how clinicians assess the right ventricles of patients with repaired congenital heart disease with residual pulmonary insufficiency. The investigators hypothesize that ultrasound enhancing agents will improve the inter-rater reliability and accuracy of various measures of right ventricular size and function, compared with cardiac MRI, thereby filling an important gap in existing methods for assessing right ventricular function. Lastly, because of the current limitations in assessing right ventricular function in this population, as a secondary aim, the investigators will also assess three-dimensional right ventricular strain -- a novel quantitative surrogate of right ventricular function.

Overall Objectives: To shift the paradigm in the assessment of right ventricular size and function by developing a protocol to assess the right ventricles in patients with repaired congenital heart disease with residual pulmonary insufficiency by integrating the use of three-dimensional echocardiography with semi-automated right ventricular analysis software with the intravenous administration of ultrasound enhancing agents.

Specific Aim 1. To compare the accuracy and inter-rater reliability of 3D echocardiography-based measurements of right ventricular end-diastolic volume, end-systolic volume, and ejection fraction, with and without contrast, with MRI derived values in patients with repaired congenital heart disease with residual pulmonary insufficiency.

Specific Aim 2. To compare the accuracy and inter-rater reliability of 3D echocardiography measurement of right ventricular strain with MRI derived right ventricular (RV) strain in patients with repaired congenital heart disease with residual pulmonary insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 11 or greater with repaired congenital heart disease and residual pulmonary insufficiency who are referred to Nemours A.I. DuPont Hospital for Children for clinically indicated cardiac MRI will be eligible for inclusion.
2. Informed written consent of parent or legal guardian.
3. Informed written assent of subject, if appropriate.

Exclusion Criteria:

1. Any patients in which Lumason is contraindicated (i.e. prior anaphylactoid reaction) will be ineligible for the clinical ultrasound and ineligible for the study.
2. History of allergic reaction to Lumason, sulfur hexafluoride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), palmitic acid)
3. Pregnant women will be excluded from the study as well since Lumason has not been studied in pregnancy.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Childrens Hospital, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinberg CR, McElhinney DB. Pulmonary valve replacement in tetralogy of Fallot. Circulation. 2014 Aug 26;130(9):795-8. doi: 10.1161/CIRCULATIONAHA.114.005551. No abstract available. PMID 25156915
- [Background] Geva T. Repaired tetralogy of Fallot: the roles of cardiovascular magnetic resonance in evaluating pathophysiology and for pulmonary valve replacement decision support. J Cardiovasc Magn Reson. 2011 Jan 20;13(1):9. doi: 10.1186/1532-429X-13-9. PMID 21251297
- [Background] Valente AM, Cook S, Festa P, Ko HH, Krishnamurthy R, Taylor AM, Warnes CA, Kreutzer J, Geva T. Multimodality imaging guidelines for patients with repaired tetralogy of fallot: a report from the AmericanSsociety of Echocardiography: developed in collaboration with the Society for Cardiovascular Magnetic Resonance and the Society for Pediatric Radiology. J Am Soc Echocardiogr. 2014 Feb;27(2):111-41. doi: 10.1016/j.echo.2013.11.009. No abstract available. PMID 24468055
- [Background] Shimada YJ, Shiota M, Siegel RJ, Shiota T. Accuracy of right ventricular volumes and function determined by three-dimensional echocardiography in comparison with magnetic resonance imaging: a meta-analysis study. J Am Soc Echocardiogr. 2010 Sep;23(9):943-53. doi: 10.1016/j.echo.2010.06.029. PMID 20797527
- [Background] Muraru D, Spadotto V, Cecchetto A, Romeo G, Aruta P, Ermacora D, Jenei C, Cucchini U, Iliceto S, Badano LP. New speckle-tracking algorithm for right ventricular volume analysis from three-dimensional echocardiographic data sets: validation with cardiac magnetic resonance and comparison with the previous analysis tool. Eur Heart J Cardiovasc Imaging. 2016 Nov;17(11):1279-1289. doi: 10.1093/ehjci/jev309. Epub 2015 Dec 8. PMID 26647080
- [Background] Laser KT, Karabiyik A, Korperich H, Horst JP, Barth P, Kececioglu D, Burchert W, DallaPozza R, Herberg U. Validation and Reference Values for Three-Dimensional Echocardiographic Right Ventricular Volumetry in Children: A Multicenter Study. J Am Soc Echocardiogr. 2018 Sep;31(9):1050-1063. doi: 10.1016/j.echo.2018.03.010. Epub 2018 Jun 19. PMID 29908725
- [Background] Medvedofsky D, Addetia K, Patel AR, Sedlmeier A, Baumann R, Mor-Avi V, Lang RM. Novel Approach to Three-Dimensional Echocardiographic Quantification of Right Ventricular Volumes and Function from Focused Views. J Am Soc Echocardiogr. 2015 Oct;28(10):1222-31. doi: 10.1016/j.echo.2015.06.013. Epub 2015 Aug 1. PMID 26237996
- [Background] Jenner J, Sorensson P, Pernow J, Caidahl K, Eriksson MJ. Contrast Enhancement and Image Quality Influence Two- and Three-dimensional Echocardiographic Determination of Left Ventricular Volumes: Comparison With Magnetic Resonance Imaging. Clin Med Insights Cardiol. 2019 Mar 5;13:1179546819831980. doi: 10.1177/1179546819831980. eCollection 2019. PMID 30858745
- [Background] van den Bosch AE, Meijboom FJ, McGhie JS, Roos-Hesselink JW, Ten Cate FJ, Roelandt JR. Enhanced visualisation of the right ventricle by contrast echocardiography in congenital heart disease. Eur J Echocardiogr. 2004 Mar;5(2):104-10. doi: 10.1016/S1525-2167(03)00048-9. PMID 15036021
- [Background] Mueller M, Rentzsch A, Hoetzer K, Raedle-Hurst T, Boettler P, Stiller B, Lemmer J, Sarikouch S, Beerbaum P, Peters B, Vogt M, Vogel M, Abdul-Khaliq H. Assessment of interventricular and right-intraventricular dyssynchrony in patients with surgically repaired tetralogy of Fallot by two-dimensional speckle tracking. Eur J Echocardiogr. 2010 Oct;11(9):786-92. doi: 10.1093/ejechocard/jeq067. Epub 2010 May 30. PMID 20513701
- [Background] Friedberg MK, Fernandes FP, Roche SL, Slorach C, Grosse-Wortmann L, Manlhiot C, Fackoury C, McCrindle BW, Mertens L, Kantor PF. Relation of right ventricular mechanics to exercise tolerance in children after tetralogy of Fallot repair. Am Heart J. 2013 Apr;165(4):551-7. doi: 10.1016/j.ahj.2012.06.029. Epub 2013 Mar 5. PMID 23537972
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Stout KK, Daniels CJ, Aboulhosn JA, Bozkurt B, Broberg CS, Colman JM, Crumb SR, Dearani JA, Fuller S, Gurvitz M, Khairy P, Landzberg MJ, Saidi A, Valente AM, Van Hare GF. 2018 AHA/ACC Guideline for the Management of Adults With Congenital Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Apr 2;73(12):1494-1563. doi: 10.1016/j.jacc.2018.08.1028. Epub 2018 Aug 16. No abstract available. PMID 30121240
- [Background] Heng EL, Gatzoulis MA, Uebing A, Sethia B, Uemura H, Smith GC, Diller GP, McCarthy KP, Ho SY, Li W, Wright P, Spadotto V, Kilner PJ, Oldershaw P, Pennell DJ, Shore DF, Babu-Narayan SV. Immediate and Midterm Cardiac Remodeling After Surgical Pulmonary Valve Replacement in Adults With Repaired Tetralogy of Fallot: A Prospective Cardiovascular Magnetic Resonance and Clinical Study. Circulation. 2017 Oct 31;136(18):1703-1713. doi: 10.1161/CIRCULATIONAHA.117.027402. PMID 29084778
- [Background] Oosterhof T, van Straten A, Vliegen HW, Meijboom FJ, van Dijk AP, Spijkerboer AM, Bouma BJ, Zwinderman AH, Hazekamp MG, de Roos A, Mulder BJ. Preoperative thresholds for pulmonary valve replacement in patients with corrected tetralogy of Fallot using cardiovascular magnetic resonance. Circulation. 2007 Jul 31;116(5):545-51. doi: 10.1161/CIRCULATIONAHA.106.659664. Epub 2007 Jul 9. PMID 17620511
- [Background] Porter TR, Mulvagh SL, Abdelmoneim SS, Becher H, Belcik JT, Bierig M, Choy J, Gaibazzi N, Gillam LD, Janardhanan R, Kutty S, Leong-Poi H, Lindner JR, Main ML, Mathias W Jr, Park MM, Senior R, Villanueva F. Clinical Applications of Ultrasonic Enhancing Agents in Echocardiography: 2018 American Society of Echocardiography Guidelines Update. J Am Soc Echocardiogr. 2018 Mar;31(3):241-274. doi: 10.1016/j.echo.2017.11.013. No abstract available. PMID 29502588
- [Background] Yusuf GT, Sellars ME, Deganello A, Cosgrove DO, Sidhu PS. Retrospective Analysis of the Safety and Cost Implications of Pediatric Contrast-Enhanced Ultrasound at a Single Center. AJR Am J Roentgenol. 2017 Feb;208(2):446-452. doi: 10.2214/AJR.16.16700. Epub 2016 Dec 13. PMID 27959665
- [Background] Piscaglia F, Bolondi L; Italian Society for Ultrasound in Medicine and Biology (SIUMB) Study Group on Ultrasound Contrast Agents. The safety of Sonovue in abdominal applications: retrospective analysis of 23188 investigations. Ultrasound Med Biol. 2006 Sep;32(9):1369-75. doi: 10.1016/j.ultrasmedbio.2006.05.031. PMID 16965977
- [Background] Kumar S, Purtell C, Peterson A, Gibbons P, Khan AM, Heitner SB. Safety profile of ultrasound enhancing agents in echocardiography. Echocardiography. 2019 Jun;36(6):1041-1044. doi: 10.1111/echo.14344. Epub 2019 Apr 30. PMID 31038768
- [Background] Yong Y, Wu D, Fernandes V, Kopelen HA, Shimoni S, Nagueh SF, Callahan JD, Bruns DE, Shaw LJ, Quinones MA, Zoghbi WA. Diagnostic accuracy and cost-effectiveness of contrast echocardiography on evaluation of cardiac function in technically very difficult patients in the intensive care unit. Am J Cardiol. 2002 Mar 15;89(6):711-8. doi: 10.1016/s0002-9149(01)02344-x. PMID 11897214
- [Background] Medvedofsky D, Mor-Avi V, Kruse E, Guile B, Ciszek B, Weinert L, Yamat M, Volpato V, Addetia K, Patel AR, Lang RM. Quantification of Right Ventricular Size and Function from Contrast-Enhanced Three-Dimensional Echocardiographic Images. J Am Soc Echocardiogr. 2017 Dec;30(12):1193-1202. doi: 10.1016/j.echo.2017.08.003. Epub 2017 Oct 17. PMID 29050828

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic Arm: The echocardiography team will perform baseline echocardiographic views of the right ventricle without contrast. The patient will receive the weight-based dose of Lumason of 0.03 mL/kg per injection, not to exceed 2.4 mL per injection per the FDA and manufacturer recommendations. Dosages and timing of administration as well as patient size and transducer type will be recorded for each patient. The total cumulative dose of Lumason from the clinical study and the research study will not exceed the maximum recommended dose by the manufacturer, 4.8 mL. A single injection will not exceed the maximal FDA-recommended dose of 2.4 mL per single injection. These echocardiographic views of the right ventricle with ultrasound enhancing agent will be compared to the measurements made without the use of ultrasound enhancing agents, and the measurements made in MRI.
  Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Injection Powder for Suspension [LUMASON]: The patient will receive the weight-based dose of Lumason of 0.03 mL/kg per injection, not to exceed 2.4 mL per injection per the FDA and manufacturer recommendations.
Period: Overall Study
Arm/Group | Diagnostic Arm
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic Arm
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Diagnosis [Count of Participants; unit: Participants] — Baseline Cardiac Diagnosis
  Participants
    Tetralogy of Fallot | 9
    Pulmonary atresia with intact ventricular septum | 4
    Pulmonary stenosis | 7
    Truncus arteriosus | 2
    Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of 3D Echocardiography Based Measurements of Right Ventricular Size Compared to MRI Derived Values.
Description: Echocardiography derived measurements of right ventricular end-diastolic volume, end-systolic volume, with and without contrast, and MRI derived values in patients with repaired congenital heart disease
Time Frame: All images were obtained on the same day of the study. MRI analysis performed by clinical reading attending. Echo analysis performed offline after completing of imaging.
Population: Two patients were unable to be analyzed for either the contrast or non-contrast group due to imaging quality and lack of complete 3D echo dataset
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Non-contrast 3D Echo: Images from non-contrast 3D echo analyzed for RV volume
- Contrast Echo: Contrast enhanced 3D echo (Lumason)
- Cardiac MRI: Measurements from clinically obtained cardiac MRI
Arm/Group | Non-contrast 3D Echo | Contrast Echo | Cardiac MRI
Number analyzed (Participants) | 21 | 17 | 24
ml
  RV End-Diastolic Volume (ml) | 187.1 (55.3) | 175.4 (53.3) | 205.0 (51.6)
  RV End-Systolic Volume (ml) | 86.0 (32.1) | 84.8 (27.5) | 100.0 (32.2)
Statistical Analysis 1: Comparison: Non-contrast 3D Echo vs Cardiac MRI; Measurements of right ventricular end-diastolic volumes were compared between two groups using an intraclass coefficient; Test type: Other; Intraclass coefficient = 0.84 — Intraclass coefficient using a two-way mixed effects model
Statistical Analysis 2: Comparison: Contrast Echo vs Cardiac MRI; [analysis description as in outcome 1, analysis 1]; Test type: Other; Intraclass coefficient = 0.77 — Intraclass coefficient using a two-way mixed effects model
Statistical Analysis 3: Comparison: Non-contrast 3D Echo vs Cardiac MRI; Measurements of right ventricular end-systolic volumes were compared between two groups using an intraclass coefficient; Test type: Other; Intraclass coefficient = 0.71 — Intraclass coefficient using a two-way mixed effects model
Statistical Analysis 4: Comparison: Contrast Echo vs Cardiac MRI; Measurements of right ventricular end-systolic volumes were compared between two groups using an intraclass coefficient; Test type: Other; Intraclass coefficient = 0.685 — Intraclass coefficient using a two-way mixed effects model

2. Primary Outcome: Accuracy of 3D Echocardiography Based Measurements of Right Ventricular Function Compared to MRI Derived Values.
Description: Echocardiography derived measurements of right ventricular ejection fraction, with and without contrast, and MRI derived values in patients with repaired congenital heart disease
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Non-contrast 3D Echo | Contrast Echo | Cardiac MRI
Number analyzed (Participants) | 21 | 17 | 24
percentage | 52 (13.8) | 52.6 (5.9) | 51.9 (6.5)
Statistical Analysis 1: Comparison: Non-contrast 3D Echo vs Cardiac MRI; Measurements of right ventricular ejection fraction were compared between non-contrast echocardiogram and cardiac MRI using an intraclass coefficient; Test type: Other; Intraclass Coefficient = 0.44 — Intraclass coefficient using a two-way mixed effects model
Statistical Analysis 2: Comparison: Contrast Echo vs Cardiac MRI; Measurements of right ventricular ejection fraction were compared between contrast echocardiogram and cardiac MRI using an intraclass coefficient; Test type: Other; Intraclass coefficient = 0.13 — Intraclass coefficient using a two-way mixed effects model

3. Primary Outcome: Inter-rater Reliability of 3D Echocardiography Based Measurements of Right Ventricular Size and Function With and Without Contrast
Description: The agreement of echocardiography derived measurements of right ventricular end-diastolic volume, end-systolic volume, and ejection fraction, with and without contrast, will be compared between the two readers using the intraclass correlation coefficient.
Time Frame: All echocardiographic images obtained on the day of the study participation. Analysis done offline.
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Comparing Echocardiographic and MRI Derived Right Ventricular Strain Measurement.
Description: 3D echocardiography measurement of right ventricular strain will be compared with MRI derived RV strain in patients with repaired congenital heart disease using an intraclass correlation coefficient.
Time Frame: Echocardiography and MRI images obtained on the day of study participation. Analysis done after image acquisition complete
Population: Images with sufficient quality were analyzed to obtain Global longitudinal strain values (expressed as a percentage)
Measure: Mean (Standard Deviation); unit: percentage strain
Groups:
- Non-contrast 3D Echo: Images from non-contrast 3D echo
- Contrast Echo: Contrast enhanced 3D echo
- Cardiac MRI: Images obtained from clinically indicated cardiac MRI
Arm/Group | Non-contrast 3D Echo | Contrast Echo | Cardiac MRI
Number analyzed (Participants) | 16 | 10 | 24
percentage strain | 23.1 (4.8) | 21.3 (5.0) | 18.1 (4.7)
Statistical Analysis 1: Comparison: Non-contrast 3D Echo vs Cardiac MRI; Test type: Other — Intraclass coefficient used to assess agreement between non-contrast echocardiographic values and cardiac MRI global longitudinal strain; Intraclass coefficient = 0.419 — Intraclass coefficient using a two-way mixed effects model
Statistical Analysis 2: Comparison: Contrast Echo vs Cardiac MRI; Test type: Other — Intraclass coefficient used to assess agreement between contrast echocardiographic values and cardiac MRI global longitudinal strain; Intraclass coefficient = 0.000 — Intraclass coefficient using a two-way mixed effects model

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | Diagnostic Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic Arm (N=25)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant reported pain which PI assessed as musculoskeletal. Resolved.

LIMITATIONS AND CAVEATS:
We acknowledge several limitations in our single-center study including the small sample size. Many patients had poor or suboptimal image quality which likely contributes to inaccuracies in calculation of RV size by echocardiography. The software used to analyze the RD echocardiography images was not designed for use with contrast enhanced echocardiograms potentially limiting the accuracy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT05186415/Prot_SAP_000.pdf